CLINICAL TRIAL: NCT03917472
Title: A 12-Month, 2-Arm, Randomized, Double-Masked, Multicenter Phase III Study Assessing the Efficacy and Safety of Brolucizumab vs. Aflibercept in Patients With Visual Impairment Due to Diabetic Macular Edema (KINGFISHER)
Brief Title: Efficacy and Safety of Brolucizumab vs Aflibercept in Patients With Visual Impairment Due to Diabetic Macular Edema
Acronym: KINGFISHER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRTH258B2305; 2019-001004-37 (EudraCT Number)
Record Dates: First submitted 2019-04-11; First posted 2019-04-17 (Actual); Results first posted 2022-04-21 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; intravitreal injection; brolucizumab; aflibercept; double-masked; Diabetic Macular edema (DME); macular edema; diabetic retinopathy
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy | interventions — brolucizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A masked evaluating investigator will be responsible for all aspects of the study except the injections and the safety assessment following the injections. An unmasked treating investigator was to perform the injections and assess patient safety following the injections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brolucizumab 6mg q4w (Experimental): Brolucizumab 6 mg/0.05 mL every 4 weeks.
  Interventions: Drug: Brolucizumab
- Aflibercept 2mg q4w (Active Comparator): Aflibercept 2mg/0.05 mL every 4 weeks
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Brolucizumab — Intravitreal injection
  Other Names: RTH258, ESBA1008
  Arms: Brolucizumab 6mg q4w
Drug: Aflibercept — Intravitreal injection
  Other Names: Eylea
  Arms: Aflibercept 2mg q4w

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of brolucizumab vs. aflibercept in the treatment of patients with visual impairment due to diabetic macular edema (DME).

DETAILED DESCRIPTION:
This study was designed as a Phase III, multi-center, randomized, double-masked, active controlled, parallel group prospective study to evaluate if brolucizumab 6 mg dosed q4w is safe and effective in the treatment of subjects with visual impairment due to diabetic macular edema (DME). Subjects who met all the inclusion and none of the exclusion criteria were randomized in a 2:1 ratio to one of two treatment arms i.e., brolucizumab 6 mg and aflibercept 2 mg. Only one eye was selected as study eye and treated with study medication.

The study included a screening period of up to 2 weeks to assess eligibility, followed by a double-masked treatment period (Day 1 to Week 48). For all subjects, the last study assessment was performed at the Week 52/end of study (EOS) visit. All subjects had study visits q4w through Week 52. The primary analysis was performed at the EOS visit (Week 52).

To ensure masking was maintained, the investigational site had both masked and unmasked staff to perform the masked and unmasked study assessments/procedures accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Patients with type 1 or type 2 diabetes mellitus (DM) and Hemoglobin A1c (HbA1c) ≤ 12% at screening.
* Study eye: Visual impairment due to DME with:

  * Best-corrected visual acuity (BCVA) score between 73 and 23 letters, inclusive, using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at an initial testing distance of 4 meters
  * DME involving the center of the macula, with Central Subfield Thickness (CSFT) ≥ 320 µm on Spectral Domain Optical Coherence Tomography (SD-OCT)

Exclusion Criteria:

* High-risk proliferative diabetic retinopathy (PDR) in the study eye
* Concomitant conditions or ocular disorders in the study eye which confound interpretation of study results, compromise visual acuity or require medical or surgical intervention
* Any active intraocular or periocular infection or active intraocular inflammation in the either eye
* Uncontrolled glaucoma in the study eye
* Presence of amblyopia, amaurosis or ocular disorders in the fellow eye with BCVA <20/200
* Use of anti-VEGF therapies, intraocular surgery or laser photocoagulation (macular or panretinal) in the study eye during the 3-month period prior to baseline
* Use of intraocular or periocular corticosteroids in the study eye during the 6-month period prior to baseline, and use of fluocinolone acetonide intravitreal (IVT) implant (Iluvien) at any time prior to baseline
* Prior investigational drugs in either eye, vitreoretinal surgery in the study eye at any time prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (85):
- United States (69):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Campbell, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Mountain View, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Poway, California
  - Novartis Investigative Site, Rancho Cordova, California
  - Novartis Investigative Site, Redlands, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Santa Barbara, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Ventura, California
  - Novartis Investigative Site, Altamonte Springs, Florida
  - Novartis Investigative Site, Deerfield Beach, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Pinellas Park, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, ‘Aiea, Hawaii
  - Novartis Investigative Site, Bloomington, Illinois
  - Novartis Investigative Site, Oak Forest, Illinois
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, New Albany, Indiana
  - Novartis Investigative Site, West Des Moines, Iowa
  - Novartis Investigative Site, Leawood, Kansas
  - Novartis Investigative Site, Lenexa, Kansas
  - Novartis Investigative Site, Hagerstown, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Royal Oak, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, Bloomfield, New Jersey
  - Novartis Investigative Site, Teaneck, New Jersey
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Hickory, North Carolina
  - Novartis Investigative Site, Southern Pines, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Dublin, Ohio
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Kingston, Pennsylvania
  - Novartis Investigative Site, Chattanooga, Tennessee
  - Novartis Investigative Site, Germantown, Tennessee
  - Novartis Investigative Site, Abilene, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Bellaire, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Harlingen, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Southlake, Texas
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Morgantown, West Virginia
  - Novartis Investigative Site, Madison, Wisconsin
- Hungary (5):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Zalaegerszeg, Zala County
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
- Novartis Investigative Site, Arecibo, Puerto Rico
- Slovakia (6):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Trebišov
  - Novartis Investigative Site, Trenčín
  - Novartis Investigative Site, Zvolen

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of the patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to criteria and process described on www.clinicalstudydatarequest.com
URL: https://clinicalstudydatarequest.com/Default.aspx

REFERENCES:
- [Derived] Singh RP, Barakat MR, Ip MS, Wykoff CC, Eichenbaum DA, Joshi S, Warrow D, Sheth VS, Stefanickova J, Kim YS, He F, Cho GE, Wang Y, Emanuelli A. Efficacy and Safety of Brolucizumab for Diabetic Macular Edema: The KINGFISHER Randomized Clinical Trial. JAMA Ophthalmol. 2023 Dec 1;141(12):1152-1160. doi: 10.1001/jamaophthalmol.2023.5248. PMID 37971723
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1085

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study centers (no. of sites): Hungary (5), Israel (5), Slovakia (7), United States (78).
  Approximately, 495 subjects were planned to be randomized. Overall, 517 subjects were randomized either to brolucizumab 6 mg q4w arm (n=346) or aflibercept 2 mg q4w arm (n=171).
Pre-assignment Details: The study included a screening period of up to 2 weeks to assess eligibility, followed by a double-masked treatment period (Day 1 to Week 48). For all subjects, the last study assessment was performed at the Week 52/end of study (EOS) visit. All subjects had study visits q4w through Week 52. The primary analysis was performed at the EOS visit (Week 52).
Period: Overall Study
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Started | 346 | 171
Completed | 311 | 156
Not Completed | 35 | 15
Not completed — Physician Decision | 4 | 0
Not completed — Adverse Event | 3 | 1
Not completed — Death | 7 | 5
Not completed — Withdrawal by Subject | 11 | 4
Not completed — Lost to Follow-up | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w | Total
Number analyzed (Participants) | 346 | 171 | 517
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 208 | 115 | 323
  >=65 years | 138 | 56 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (10.59) | 60.2 (9.31) | 60.7 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 66 | 218
  Male | 194 | 105 | 299
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 14 | 7 | 21
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 40 | 15 | 55
  White | 288 | 145 | 433
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best-corrected Visual Acuity (BCVA) at Week 52
Description: BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score of 73 to 23 (per the inclusion criteria) (approximate Snellen equivalent of 20/40 to 20/320) in the study eye were included.
  Min and max possible scores are 0-100 respectively. A higher score represents better functioning.
  Last observation carried forward (LOCF) was used for the imputation of missing values.
Time Frame: Baseline, Week 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 346 | 171
Scores on a scale | 12.2 [11.2 to 13.2] | 11.0 [9.6 to 12.4]
Statistical Analysis 1: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; Test type: Superiority — (1-sided); p = 0.099, ANOVA; LS mean difference = 1.1, 95% CI 2-sided [-0.6 to 2.9], Standard Error of Mean 0.89
Statistical Analysis 2: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; Test type: Non-Inferiority — (4-letter margin) (1-sided); p < 0.001, ANOVA

2. Secondary Outcome: Change From Baseline in Central Subfield Thickness (CSFT) at Each Post-baseline Visit
Description: Central Subfield Thickness assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center.
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: μm
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 346 | 171
μm
  Week 4 | -146.9 [-157.9 to -136.0] | -119.5 [-135.1 to -103.9]
  Week 8 | -174.4 [-185.3 to -163.4] | -144.1 [-159.7 to -128.5]
  Week 12 | -191.3 [-201.8 to -180.8] | -156.7 [-171.7 to -141.8]
  Week 16 | -200.5 [-211.0 to -189.9] | -162.4 [-177.4 to -147.4]
  Week 20 | -209.5 [-219.6 to -199.4] | -168.7 [-183.1 to -154.2]
  Week 24 | -217.5 [-227.3 to -207.6] | -178.8 [-192.8 to -164.7]
  Week 28 | -222.4 [-232.5 to -212.4] | -183.6 [-197.8 to -169.3]
  Week 32 | -227.2 [-237.2 to -217.1] | -185.9 [-200.2 to -171.6]
  Week 36 | -229.7 [-240.1 to -219.3] | -186.7 [-201.5 to -172.0]
  Week 40 | -233.6 [-243.7 to -223.6] | -188.4 [-202.6 to -174.1]
  Week 44 | -237.5 [-247.4 to -227.5] | -188.1 [-202.3 to -173.9]
  Week 48 | -237.7 [-247.7 to -227.6] | -192.0 [-206.4 to -177.7]
  Week 52 | -237.8 [-247.9 to -227.7] | -196.5 [-210.8 to -182.1]
Statistical Analysis 1: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; Test type: Superiority — (1-sided); Week 52; p < 0.001, ANOVA; LS mean difference = -41.4, 95% CI 2-sided [-58.9 to -23.8], Standard Error of Mean 8.94

3. Secondary Outcome: Number and Percentage of Participants With Fluid-free Macula in the Study Eye at Each Post-baseline Visit
Description: Subretinal Fluid (SRF) and Intraretinal Fluid (IRF) status in the central subfield: proportion of subjects with simultaneous absence of SRF and IRF in the study eye by visit. Events and censoring after 52 weeks are included in week 52 row.
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF).
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 346 | 171
Participants
  Week 4 | 23 | 4
  Week 8 | 31 | 4
  Week 12 | 38 | 10
  Week 16 | 48 | 11
  Week 20 | 54 | 9
  Week 24 | 84 | 19
  Week 28 | 65 | 13
  Week 32 | 76 | 17
  Week 36 | 91 | 21
  Week 40 | 96 | 23
  Week 44 | 96 | 20
  week 48 | 92 | 23
  Week 52 | 144 | 38
Statistical Analysis 1: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; Test type: Superiority — (1-sided) Week 52; p < 0.001, Clopper-Pearson exact method; Difference - % = 20.0, 95% CI 2-sided [12.5 to 28.6]

4. Secondary Outcome: Number and Percentage of Participants With Absence of Diabetic Macular Edema (DME) (CSFT < 280 μm) at Each Post-baseline Visit for the Study Eye
Description: as for outcome 2
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 346 | 171
Participants
  Week 4 | 61 | 9
  Week 8 | 93 | 24
  Week 12 | 124 | 33
  Week 16 | 147 | 42
  Week 20 | 167 | 47
  Week 24 | 177 | 52
  Week 28 | 186 | 57
  Week 32 | 195 | 62
  Week 36 | 206 | 63
  Week 40 | 211 | 65
  Week 44 | 216 | 69
  Week 48 | 222 | 68
  Week 52 | 229 | 71

5. Secondary Outcome: Time to First Fluid-free Macula - Time-to-first Absence of Subretinal Fluid (SRF) and Intraretinal Fluid (IRF) in the Study Eye - Number of Subjects With Absence of SRF / IRF and Number of Subjects Censored by Visit
Description: Central Subfield Thickness Assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center. Fluid status assessments after start of alternative DME treatment in the study eye are censored. Time to first fluid-free macula analysis is based on the subset of subjects with fluid present at baseline and at least one post-baseline assessment. Time (week) was calculated by (study day / 7). Events and censoring after 52 weeks were included in week 52 row.
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and 52
Population: Full Analysis Set. Time to first fluid-free macula analysis is based on the subset of subjects with fluid present at baseline and at least one post-baseline assessment.
Measure: Number; unit: Participants
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 344 | 170
Participants
  Number of subjects with absence of SRF / IRF at Week 0 (n=344,170) | 0 | 0
  Number of subjects with absence of SRF / IRF at Week 4 (n=344,170) | 6 | 1
  Number of subjects with absence of SRF / IRF at Week 8 (n=335,168): number analyzed (Participants) | 335 | 168
  Number of subjects with absence of SRF / IRF at Week 8 (n=335,168) | 18 | 3
  Number of subjects with absence of SRF / IRF at Week 12 (n=314, 165): number analyzed (Participants) | 314 | 165
  Number of subjects with absence of SRF / IRF at Week 12 (n=314, 165) | 13 | 2
  Number of subjects with absence of SRF / IRF at Week 16 (n=297, 161): number analyzed (Participants) | 297 | 161
  Number of subjects with absence of SRF / IRF at Week 16 (n=297, 161) | 17 | 4
  Number of subjects with absence of SRF / IRF at Week 20 (n=277, 156): number analyzed (Participants) | 277 | 156
  Number of subjects with absence of SRF / IRF at Week 20 (n=277, 156) | 8 | 6
  Number of subjects with absence of SRF / IRF at Week 24 (n=265,150): number analyzed (Participants) | 265 | 150
  Number of subjects with absence of SRF / IRF at Week 24 (n=265,150) | 16 | 2
  Number of subjects with absence of SRF / IRF at Week 28 (n=246,146): number analyzed (Participants) | 246 | 146
  Number of subjects with absence of SRF / IRF at Week 28 (n=246,146) | 18 | 7
  Number of subjects with absence of SRF / IRF at Week 32 (n=224,139): number analyzed (Participants) | 224 | 139
  Number of subjects with absence of SRF / IRF at Week 32 (n=224,139) | 3 | 1
  Number of subjects with absence of SRF / IRF at Week 36 (n=220,138): number analyzed (Participants) | 220 | 138
  Number of subjects with absence of SRF / IRF at Week 36 (n=220,138) | 8 | 2
  Number of subjects with absence of SRF / IRF at Week 40 (n=211, 134): number analyzed (Participants) | 211 | 134
  Number of subjects with absence of SRF / IRF at Week 40 (n=211, 134) | 16 | 4
  Number of subjects with absence of SRF / IRF at Week 44 (194, 129): number analyzed (Participants) | 194 | 129
  Number of subjects with absence of SRF / IRF at Week 44 (194, 129) | 11 | 2
  Number of subjects with absence of SRF / IRF at Week 48 (n=181, 125): number analyzed (Participants) | 181 | 125
  Number of subjects with absence of SRF / IRF at Week 48 (n=181, 125) | 3 | 0
  Number of subjects with absence of SRF / IRF at Week 52 (n=177, 122): number analyzed (Participants) | 177 | 122
  Number of subjects with absence of SRF / IRF at Week 52 (n=177, 122) | 30 | 12
  Number of subjects censored at Week 0 (n=344, 170) | 0 | 0
  Number of subjects censored at Week 4 (n-344, 170) | 3 | 1
  Number of subjects censored at Week 8 (n=335,168): number analyzed (Participants) | 335 | 168
  Number of subjects censored at Week 8 (n=335,168) | 3 | 0
  Number of subjects censored at Week 12 (n=314, 165): number analyzed (Participants) | 314 | 165
  Number of subjects censored at Week 12 (n=314, 165) | 4 | 2
  Number of subjects censored at Week 16 (n=297, 161): number analyzed (Participants) | 297 | 161
  Number of subjects censored at Week 16 (n=297, 161) | 3 | 1
  Number of subjects censored at Week 20 (n=277, 156): number analyzed (Participants) | 277 | 156
  Number of subjects censored at Week 20 (n=277, 156) | 4 | 0
  Number of subjects censored at Week 24 (n=265, 150): number analyzed (Participants) | 265 | 150
  Number of subjects censored at Week 24 (n=265, 150) | 3 | 2
  Number of subjects censored at Week 28 (n=246, 146): number analyzed (Participants) | 246 | 146
  Number of subjects censored at Week 28 (n=246, 146) | 4 | 0
  Number of subjects censored at Week 32 (n=224,139): number analyzed (Participants) | 224 | 139
  Number of subjects censored at Week 32 (n=224,139) | 1 | 0
  Number of subjects censored at Week 36 (220, 138): number analyzed (Participants) | 220 | 138
  Number of subjects censored at Week 36 (220, 138) | 1 | 2
  Number of subjects censored at Week 40 (n=211,134): number analyzed (Participants) | 211 | 134
  Number of subjects censored at Week 40 (n=211,134) | 1 | 1
  Number of subjects censored at Week 44 (n=194,129): number analyzed (Participants) | 194 | 129
  Number of subjects censored at Week 44 (n=194,129) | 2 | 2
  Number of subjects censored at Week 48 (n=181, 125): number analyzed (Participants) | 181 | 125
  Number of subjects censored at Week 48 (n=181, 125) | 1 | 3
  Number of subjects censored at Week 52 (n=177, 122): number analyzed (Participants) | 177 | 122
  Number of subjects censored at Week 52 (n=177, 122) | 147 | 110

6. Secondary Outcome: Time to First Fluid-free Macula - Time-to-first Absence of Subretinal Fluid (SRF) and Intraretinal Fluid (IRF) in the Study Eye - Kaplan-Meier Analysis - Probability of Absence of SRF/IRF by Visit
Description: as for outcome 5
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Probability of absence of SRF/IRF
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 344 | 170
Probability of absence of SRF/IRF
  Probability of absence of SRF/IRF at Week 0 (n=344,170) | 0.000 [NA to NA] — CIs are not applicable for probability = 0. | 0.000 [NA to NA] — CIs are not applicable for probability = 0.
  Probability of absence of SRF/IRF at Week 4 (n=344,170) | 0.018 [0.007 to 0.036] | 0.006 [0.001 to 0.030]
  Probability of absence of SRF/IRF at Week 8 (n=335,168): number analyzed (Participants) | 335 | 168
  Probability of absence of SRF/IRF at Week 8 (n=335,168) | 0.071 [0.047 to 0.101] | 0.024 [0.008 to 0.056]
  Probability of absence of SRF/IRF at Week 12 (n=314, 165): number analyzed (Participants) | 314 | 165
  Probability of absence of SRF/IRF at Week 12 (n=314, 165) | 0.109 [0.079 to 0.145] | 0.036 [0.015 to 0.072]
  Probability of absence of SRF/IRF at Week 16 (n=297, 161): number analyzed (Participants) | 297 | 161
  Probability of absence of SRF/IRF at Week 16 (n=297, 161) | 0.161 [0.124 to 0.202] | 0.060 [0.030 to 0.103]
  Probability of absence of SRF/IRF at Week 20 (n=277, 156): number analyzed (Participants) | 277 | 156
  Probability of absence of SRF/IRF at Week 20 (n=277, 156) | 0.185 [0.145 to 0.228] | 0.096 [0.057 to 0.146]
  Probability of absence of SRF/IRF at Week 24 (n=265,150): number analyzed (Participants) | 265 | 150
  Probability of absence of SRF/IRF at Week 24 (n=265,150) | 0.234 [0.190 to 0.281] | 0.108 [0.067 to 0.161]
  Probability of absence of SRF/IRF at Week 28 (n=246,146): number analyzed (Participants) | 246 | 146
  Probability of absence of SRF/IRF at Week 28 (n=246,146) | 0.291 [0.243 to 0.341] | 0.151 [0.101 to 0.210]
  Probability of absence of SRF/IRF at Week 32 (n=224,139): number analyzed (Participants) | 224 | 139
  Probability of absence of SRF/IRF at Week 32 (n=224,139) | 0.300 [0.252 to 0.351] | 0.157 [0.106 to 0.217]
  Probability of absence of SRF/IRF at Week 36 (n=220,138): number analyzed (Participants) | 220 | 138
  Probability of absence of SRF/IRF at Week 36 (n=220,138) | 0.326 [0.275 to 0.377] | 0.169 [0.116 to 0.230]
  Probability of absence of SRF/IRF at Week 40 (n=211, 134): number analyzed (Participants) | 211 | 134
  Probability of absence of SRF/IRF at Week 40 (n=211, 134) | 0.377 [0.324 to 0.430] | 0.194 [0.137 to 0.258]
  Probability of absence of SRF/IRF at Week 44 (194, 129): number analyzed (Participants) | 194 | 129
  Probability of absence of SRF/IRF at Week 44 (194, 129) | 0.412 [0.358 to 0.466] | 0.206 [0.148 to 0.271]
  Probability of absence of SRF/IRF at Week 48 (n=181, 125): number analyzed (Participants) | 181 | 125
  Probability of absence of SRF/IRF at Week 48 (n=181, 125) | 0.422 [0.368 to 0.476] | 0.206 [0.148 to 0.271]
  Probability of absence of SRF/IRF at Week 52 (n=177, 122): number analyzed (Participants) | 177 | 122
  Probability of absence of SRF/IRF at Week 52 (n=177, 122) | 0.653 [0.540 to 0.745] | 0.328 [0.234 to 0.426]

7. Secondary Outcome: Time to First Absence of Diabetic Macular Edema (DME) (CSFT < 280 μm) in the Study Eye at Each Post-baseline Visit - Number of Subjects With Probability of Absence of DME and Number Censored by Visit
Description: Central Subfield Thickness Assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center. CSFT assessments after start of alternative DME treatment in the study eye are censored. Time to first absence of DME based on subjects with valid baseline and at least one post-baseline CSFT assessment. Time (week) was calculated by (study day / 7). Events and censoring after 52 weeks were included in week 52 row.
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and 52
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 346 | 171
Participants
  Number of subjects with Probability of absence of DME at Week 0 (n=346,171) | 0 | 0
  Number of subjects with Probability of absence of DME at Week 4 (n=346,171) | 14 | 1
  Number of subjects with Probability of absence of DME at Week 8 (n=329,169): number analyzed (Participants) | 329 | 169
  Number of subjects with Probability of absence of DME at Week 8 (n=329,169) | 54 | 12
  Number of subjects with Probability of absence of DME at Week 12 (n=272, 157): number analyzed (Participants) | 272 | 157
  Number of subjects with Probability of absence of DME at Week 12 (n=272, 157) | 32 | 13
  Number of subjects with Probability of absence of DME at Week 16 (n=239, 142): number analyzed (Participants) | 239 | 142
  Number of subjects with Probability of absence of DME at Week 16 (n=239, 142) | 33 | 11
  Number of subjects with Probability of absence of DME at Week 20 (n=204, 130): number analyzed (Participants) | 204 | 130
  Number of subjects with Probability of absence of DME at Week 20 (n=204, 130) | 26 | 10
  Number of subjects with Probability of absence of DME at Week 24 (n=174,120): number analyzed (Participants) | 174 | 120
  Number of subjects with Probability of absence of DME at Week 24 (n=174,120) | 12 | 4
  Number of subjects with Probability of absence of DME at Week 28 (n=161,115): number analyzed (Participants) | 161 | 115
  Number of subjects with Probability of absence of DME at Week 28 (n=161,115) | 13 | 7
  Number of subjects with Probability of absence of DME at Week 32 (n=146,107): number analyzed (Participants) | 146 | 107
  Number of subjects with Probability of absence of DME at Week 32 (n=146,107) | 9 | 5
  Number of subjects with Probability of absence of DME at Week 36 (n=135,102): number analyzed (Participants) | 135 | 102
  Number of subjects with Probability of absence of DME at Week 36 (n=135,102) | 10 | 2
  Number of subjects with Probability of absence of DME at Week 40 (n=125, 98): number analyzed (Participants) | 125 | 98
  Number of subjects with Probability of absence of DME at Week 40 (n=125, 98) | 7 | 1
  Number of subjects with Probability of absence of DME at Week 44 (117, 96): number analyzed (Participants) | 117 | 96
  Number of subjects with Probability of absence of DME at Week 44 (117, 96) | 11 | 2
  Number of subjects with Probability of absence of DME at Week 48 (n=106, 92): number analyzed (Participants) | 106 | 92
  Number of subjects with Probability of absence of DME at Week 48 (n=106, 92) | 6 | 3
  Number of subjects with Probability of absence of DME at Week 52 (n=99, 88): number analyzed (Participants) | 99 | 88
  Number of subjects with Probability of absence of DME at Week 52 (n=99, 88) | 13 | 4
  Number censored at Week 0 (n=346,171) | 0 | 0
  Number censored at Week 4 (n=346,171) | 3 | 1
  Number censored at Week 8 (n=329,169): number analyzed (Participants) | 329 | 169
  Number censored at Week 8 (n=329,169) | 3 | 0
  Number censored at Week 12 (n=272, 157): number analyzed (Participants) | 272 | 157
  Number censored at Week 12 (n=272, 157) | 1 | 2
  Number censored at Week 16 (n=239, 142): number analyzed (Participants) | 239 | 142
  Number censored at Week 16 (n=239, 142) | 2 | 1
  Number censored at Week 20 (n=204, 130): number analyzed (Participants) | 204 | 130
  Number censored at Week 20 (n=204, 130) | 4 | 0
  Number censored at Week 24 (n=174,120): number analyzed (Participants) | 174 | 120
  Number censored at Week 24 (n=174,120) | 1 | 1
  Number censored at Week 28 (n=161,115): number analyzed (Participants) | 161 | 115
  Number censored at Week 28 (n=161,115) | 2 | 1
  Number censored at Week 32 (n=146,107): number analyzed (Participants) | 146 | 107
  Number censored at Week 32 (n=146,107) | 2 | 0
  Number censored at Week 36 (n=135,102): number analyzed (Participants) | 135 | 102
  Number censored at Week 36 (n=135,102) | 0 | 2
  Number censored at Week 40 (n=125, 98): number analyzed (Participants) | 125 | 98
  Number censored at Week 40 (n=125, 98) | 1 | 1
  Number censored at Week 44 (117, 96): number analyzed (Participants) | 117 | 96
  Number censored at Week 44 (117, 96) | 0 | 2
  Number censored at Week 48 (n=106, 92): number analyzed (Participants) | 106 | 92
  Number censored at Week 48 (n=106, 92) | 1 | 1
  Number censored at Week 52 (n=99, 88): number analyzed (Participants) | 99 | 88
  Number censored at Week 52 (n=99, 88) | 86 | 84

8. Secondary Outcome: Time to First Absence of Diabetic Macular Edema (DME) (CSFT < 280 μm) in the Study Eye at Each Post-baseline Visit - Kaplan-Meier Analysis - Probability of Absence of DME by Visit
Description: as for outcome 7
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and 52
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Probability of absence of DME
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 346 | 171
Probability of absence of DME
  Probability of absence of DME at Week 0 (n=346,171) | 0.000 [NA to NA] — CIs are not applicable when the probability = 0. | 0.000 [NA to NA] — CIs are not applicable when the probability = 0.
  Probability of absence of DME at Week 4 (n=346,171) | 0.041 [0.023 to 0.066] | 0.006 [0.001 to 0.030]
  Probability of absence of DME at Week 8 (n=329,169): number analyzed (Participants) | 329 | 169
  Probability of absence of DME at Week 8 (n=329,169) | 0.199 [0.158 to 0.243] | 0.076 [0.043 to 0.123]
  Probability of absence of DME at Week 12 (n=272, 157): number analyzed (Participants) | 272 | 157
  Probability of absence of DME at Week 12 (n=272, 157) | 0.293 [0.246 to 0.342] | 0.153 [0.104 to 0.212]
  Probability of absence of DME at Week 16 (n=239, 142): number analyzed (Participants) | 239 | 142
  Probability of absence of DME at Week 16 (n=239, 142) | 0.391 [0.339 to 0.443] | 0.219 [0.160 to 0.284]
  Probability of absence of DME at Week 20 (n=204, 130): number analyzed (Participants) | 204 | 130
  Probability of absence of DME at Week 20 (n=204, 130) | 0.470 [0.416 to 0.522] | 0.279 [0.213 to 0.348]
  Probability of absence of DME at Week 24 (n=174,120): number analyzed (Participants) | 174 | 120
  Probability of absence of DME at Week 24 (n=174,120) | 0.506 [0.452 to 0.559] | 0.303 [0.235 to 0.374]
  Probability of absence of DME at Week 28 (n=161,115): number analyzed (Participants) | 161 | 115
  Probability of absence of DME at Week 28 (n=161,115) | 0.547 [0.491 to 0.598] | 0.346 [0.274 to 0.418]
  Probability of absence of DME at Week 32 (n=146,107): number analyzed (Participants) | 146 | 107
  Probability of absence of DME at Week 32 (n=146,107) | 0.575 [0.520 to 0.626] | 0.376 [0.303 to 0.450]
  Probability of absence of DMEE at Week 36 (n=135,102): number analyzed (Participants) | 135 | 102
  Probability of absence of DMEE at Week 36 (n=135,102) | 0.606 [0.551 to 0.657] | 0.389 [0.314 to 0.462]
  Probability of absence of DME at Week 40 (n=125, 98): number analyzed (Participants) | 125 | 98
  Probability of absence of DME at Week 40 (n=125, 98) | 0.628 [0.574 to 0.678] | 0.395 [0.320 to 0.468]
  Probability of absence of DME at Week 44 (117, 96): number analyzed (Participants) | 117 | 96
  Probability of absence of DME at Week 44 (117, 96) | 0.663 [0.609 to 0.712] | 0.408 [0.332 to 0.482]
  Probability of absence of DME at Week 48 (n=106, 92): number analyzed (Participants) | 106 | 92
  Probability of absence of DME at Week 48 (n=106, 92) | 0.682 [0.629 to 0.730] | 0.427 [0.351 to 0.501]
  Probability of absence of DME at Week 52 (n=99, 88): number analyzed (Participants) | 99 | 88
  Probability of absence of DME at Week 52 (n=99, 88) | 0.866 [0.302 to 0.983] | 0.516 [0.357 to 0.654]

9. Secondary Outcome: Best Corrected Visual Acuity (Letters Read): Change From Baseline in Best-corrected Visual Acuity (BCVA) at Each Post-baseline Visit for the Study Eye
Description: BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score of 73 to 23 (per the inclusion criteria) (approximate Snellen equivalent of 20/40 to 20/320) in the study eye were included.
  Min and max possible scores are 0-100 respectively. A higher score represents better functioning.
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 346 | 171
scores on a scale
  Week 4 | 5.7 [5.1 to 6.4] | 5.4 [4.5 to 6.4]
  Week 8 | 7.7 [6.9 to 8.5] | 7.4 [6.4 to 8.5]
  Week 12 | 9.1 [8.3 to 9.9] | 8.0 [6.9 to 9.1]
  Week 16 | 9.6 [8.8 to 10.4] | 8.5 [7.3 to 9.7]
  Week 20 | 10.2 [9.3 to 11.1] | 9.2 [7.9 to 10.5]
  Week 24 | 10.7 [9.8 to 11.6] | 9.6 [8.3 to 10.9]
  Week 28 | 10.9 [10.0 to 11.8] | 10.7 [9.3 to 12.0]
  Week 32 | 11.5 [10.6 to 12.5] | 10.5 [9.2 to 11.9]
  Week 36 | 11.6 [10.6 to 12.6] | 10.8 [9.4 to 12.2]
  Week 40 | 11.7 [10.7 to 12.6] | 10.7 [9.4 to 12.1]
  Week 44 | 12.0 [11.0 to 13.0] | 10.6 [9.2 to 12.0]
  Week 48 | 12.2 [11.2 to 13.2] | 10.7 [9.3 to 12.1]
  Week 52 | 12.2 [11.2 to 13.2] | 11.0 [9.6 to 12.4]

10. Secondary Outcome: Gain in Best-corrected Visual Acuity (BCVA) (Letters Read): Number (%) of Subjects Who Gained ≥ 5, 10, or 15 Letters in BCVA From Baseline or Reached BCVA ≥ 84 Letters in the Study Eye at Week 52
Description: as for outcome 9
Time Frame: Baseline, Week 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 346 | 171
Participants
  ≥ 5 letters gain from baseline or BCVA ≥ 84 letters at Week 52 | 286 [78.2 to 86.5] | 127 [67.0 to 80.6]
  ≥ 10 letters gain from baseline or BCVA ≥ 84 letters at Week 52 | 211 [55.6 to 66.2] | 95 [47.8 to 63.1]
  ≥ 15 letters gain from baseline or BCVA ≥ 84 letters at Week 52 | 151 [38.3 to 49.0] | 69 [32.9 to 48.1]
Statistical Analysis 1: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; ≥ 5 letters gain from baseline or BCVA ≥ 84 letters at Week 52; Test type: Other — Descriptive; Clopper-Pearson exact method; Difference - % = 9.3, 95% CI 2-sided [1.7 to 17.0]
Statistical Analysis 2: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; ≥ 10 letters gain from baseline or BCVA ≥ 84 letters at Week 52; Test type: Other — Descriptive; Clopper-Pearson exact method; Difference - % = 7.7, 95% CI 2-sided [-1.5 to 17.0]
Statistical Analysis 3: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; ≥ 15 letters gain from baseline or BCVA ≥ 84 letters at Week 52; Test type: Other — Descriptive; Clopper-Pearson exact method; Difference - % = 5.5, 95% CI 2-sided [-2.7 to 14.3]

11. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Proportion of Subjects With >=2-step Improvement From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye
Description: The Diabetic Retinopathy Disease Severity Scale measures the 5 levels of diabetic retinopathy - none, mild, moderate, severe, and proliferative.
  Severity of Diabetic retinopathy was evaluated using the ETDRS DRSS score assessed by the Central Reading Center based on color fundus photography images in the study eye. When the ETDRS-DR severities were evaluable, they were categorized on the original scale with scores varying from 10 (DR absent) to 85 (very advanced PDR). All DRSS values were then converted into a 12-level scale, allowing the derivation of the ≥2-step and ≥3-step change from baseline for each post-baseline assessment".
  A lower score represents better functioning.
  Subjects who had full/partial panretinal photocoagulation or local photocoagulation for new vessel (DRSS score 60) at any visit were excluded.
  DRSS scores after start of alternative DME treatment in the study eye are censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: Baseline, Weeks 12, 24 and 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF). Subjects who had full/partial panretinal photocoagulation or local photocoagulation for new vessel (DRSS score 60) at any visit were excluded from analysis.
  DRSS scores after start of alternative DME treatment in the study eye are censored and replaced by the last value prior to start of this alternative treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 221 | 118
Participants
  Week 12 | 56 | 21
  Week 24 | 82 | 38
  Week 52 | 95 | 45
Statistical Analysis 1: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; Test type: Other — descriptive; week 12; Clopper-Pearson exact method; Difference - % = 8.3, 95% CI 2-sided [0.2 to 16.5]
Statistical Analysis 2: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; Test type: Other — descriptive; week 24; Clopper-Pearson exact method; Difference - % = 6.0, 95% CI 2-sided [-3.0 to 14.9]
Statistical Analysis 3: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; Test type: Non-Inferiority — (10% margin); week 52; p = 0.002, Clopper-Pearson exact method — (10% margin) (1-sided); Difference - % = 6.0, 95% CI 2-sided [-3.9 to 16.1]

12. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Proportion of Subjects With >=3-step Improvement From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye
Description: as for outcome 11
Time Frame: Baseline, Weeks 12, 24 and 52
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 221 | 118
Participants
  Week 12 | 18 | 8
  Week 24 | 33 | 16
  Week 52 | 40 | 18
Statistical Analysis 1: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; Test type: Other — descriptive; week 12; Clopper-Pearson exact method; Difference - % = 2.0, 95% CI 2-sided [-2.5 to 6.6]
Statistical Analysis 2: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; Test type: Other — descriptive; week 24; Clopper-Pearson exact method; Difference - % = 2.4, 95% CI 2-sided [-3.0 to 7.7]
Statistical Analysis 3: Comparison: Brolucizumab 6mg q4w vs Aflibercept 2mg q4w; Test type: Other — descriptive; week 52; Clopper-Pearson exact method; Difference - % = 3.9, 95% CI 2-sided [-2.0 to 9.8]

13. Secondary Outcome: Anti-Drug Antibody (ADA): Frequency Distribution of Pre-existing ADA Status in the Brolucizumab Arm
Time Frame: Baseline
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6mg q4w
Number analyzed (Participants) | 342
Participants
  Negative | 112
  Positive | 230

14. Secondary Outcome: Ocular AEs (Greater Than or Equal to 2% in Any Treatment Arm) by Preferred Term in the Study Eye
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 52 weeks.
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 346 | 171
Participants
  Number of subjects with at least one AE | 105 | 59
  Vitreous detachment | 10 | 7
  Cataract | 9 | 6
  Conjunctival haemorrhage | 9 | 7
  Punctate keratitis | 9 | 2
  Uveitis | 8 | 1
  Vitreous floaters | 8 | 5
  Dry eye | 7 | 4
  Eye pain | 6 | 5
  Corneal abrasion | 0 | 5
  Diabetic retinal oedema | 0 | 4

15. Secondary Outcome: Number of Subjects With Non-ocular AEs (Greater Than or Equal to 2% in Any Treatment Arm)
Time Frame: as for outcome 14
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6mg q4w | Aflibercept 2mg q4w
Number analyzed (Participants) | 346 | 171
Participants | 209 | 96

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 52 weeks.
Groups:
- Brolucizumab 6mg: Brolucizumab 6mg
- Aflibercept 2mg: Aflibercept 2mg
- Overall: Overall
Arm/Group | Brolucizumab 6mg | Aflibercept 2mg | Overall
All-Cause Mortality (participants affected / at risk) | 7/346 | 5/171 | 12/517
Serious Adverse Events (participants affected / at risk) | 74/346 | 36/171 | 110/517
Other Adverse Events (participants affected / at risk) | 144/346 | 92/171 | 236/517
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=346) | Aflibercept 2mg (N=171) | Overall (N=517)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 2
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 2 | 0 | 2
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 3 | 1 | 4
Cardiac failure congestive (Cardiac disorders) | 4 | 0 | 4
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 1 | 4
Left ventricular failure (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 3 | 1 | 4
Myocardial ischaemia (Cardiac disorders) | 2 | 1 | 3
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Cataract - Fellow eye (Eye disorders) | 0 | 1 | 1
Cataract subcapsular - Study eye (Eye disorders) | 1 | 0 | 1
Diabetic retinopathy - Fellow eye (Eye disorders) | 1 | 0 | 1
Retinal vasculitis - Study eye (Eye disorders) | 1 | 0 | 1
Vitreous haemorrhage - Fellow eye (Eye disorders) | 2 | 0 | 2
Vitreous haemorrhage - Study eye (Eye disorders) | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Peripheral swelling (General disorders) | 1 | 0 | 1
Sudden death (General disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 1
Abscess bacterial (Infections and infestations) | 1 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 1
Bronchitis viral (Infections and infestations) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 8 | 1 | 9
COVID-19 pneumonia (Infections and infestations) | 4 | 0 | 4
Cellulitis (Infections and infestations) | 3 | 0 | 3
Chest wall abscess (Infections and infestations) | 1 | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 1
Diabetic foot infection (Infections and infestations) | 1 | 2 | 3
Diabetic gangrene (Infections and infestations) | 0 | 1 | 1
Gangrene (Infections and infestations) | 2 | 1 | 3
Kidney infection (Infections and infestations) | 1 | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 3 | 2 | 5
Pneumonia (Infections and infestations) | 3 | 2 | 5
Sepsis (Infections and infestations) | 2 | 1 | 3
Septic shock (Infections and infestations) | 1 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 1
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Cataract operation complication - Fellow eye (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 1
Blood potassium increased (Investigations) | 1 | 0 | 1
Troponin increased (Investigations) | 1 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 6 | 6 | 12
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 2
Lacunar stroke (Nervous system disorders) | 1 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 4 | 1 | 5
Chronic kidney disease (Renal and urinary disorders) | 3 | 0 | 3
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1
Renal mass (Renal and urinary disorders) | 1 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Diabetic wound (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Extremity necrosis (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 2 | 3
Hypertensive emergency (Vascular disorders) | 1 | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=346) | Aflibercept 2mg (N=171) | Overall (N=517)
Anaemia (Blood and lymphatic system disorders) | 8 | 4 | 12
Cataract - Fellow eye (Eye disorders) | 6 | 4 | 10
Cataract - Study eye (Eye disorders) | 9 | 6 | 15
Conjunctival haemorrhage - Fellow eye (Eye disorders) | 4 | 5 | 9
Conjunctival haemorrhage - Study eye (Eye disorders) | 9 | 7 | 16
Diabetic retinal oedema - Fellow eye (Eye disorders) | 10 | 7 | 17
Diabetic retinal oedema - Study eye (Eye disorders) | 0 | 4 | 4
Dry eye - Fellow eye (Eye disorders) | 6 | 6 | 12
Dry eye - Study eye (Eye disorders) | 7 | 4 | 11
Eye pain - Fellow eye (Eye disorders) | 3 | 4 | 7
Eye pain - Study eye (Eye disorders) | 6 | 5 | 11
Punctate keratitis - Study eye (Eye disorders) | 9 | 2 | 11
Uveitis - Study eye (Eye disorders) | 8 | 1 | 9
Vitreous detachment - Study eye (Eye disorders) | 10 | 7 | 17
Vitreous floaters - Study eye (Eye disorders) | 8 | 5 | 13
Vitreous haemorrhage - Fellow eye (Eye disorders) | 10 | 4 | 14
Nausea (Gastrointestinal disorders) | 3 | 4 | 7
Oedema peripheral (General disorders) | 3 | 4 | 7
Pyrexia (General disorders) | 4 | 4 | 8
COVID-19 (Infections and infestations) | 11 | 11 | 22
Cellulitis (Infections and infestations) | 7 | 4 | 11
Influenza (Infections and infestations) | 2 | 4 | 6
Nasopharyngitis (Infections and infestations) | 8 | 6 | 14
Urinary tract infection (Infections and infestations) | 11 | 2 | 13
Corneal abrasion - Study eye (Injury, poisoning and procedural complications) | 0 | 5 | 5
Fall (Injury, poisoning and procedural complications) | 9 | 4 | 13
Blood creatinine increased (Investigations) | 4 | 7 | 11
Blood pressure increased (Investigations) | 7 | 5 | 12
Diabetes mellitus (Metabolism and nutrition disorders) | 7 | 0 | 7
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 | 4 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 7
Headache (Nervous system disorders) | 3 | 7 | 10
Acute kidney injury (Renal and urinary disorders) | 8 | 4 | 12
Chronic kidney disease (Renal and urinary disorders) | 8 | 4 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 12
Hypertension (Vascular disorders) | 18 | 13 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03917472/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT03917472/SAP_001.pdf